CLINICAL TRIAL: NCT04934306
Title: Normative Nasalance Scores for Native French-speaking Children
Brief Title: Nasalance Scores for Normal-speaking French Children
Acronym: NONAFRA2022
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210445; 2021-A00452-39 (Other: IDRCB)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Resonance Disorder
Keywords: Nasometer; Nasometry; Nasalance scores; Velopharyngeal dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients without cleft: Patients without developmental speech disorder (including articulation disorder) or hearing impairment
  Interventions: Other: Nasometry
- Patients with a cleft: Patients with a hard and/or soft palate cleft and for whom the perceptual speech-language pathology evaluation revealed a velopharyngeal insufficiency
  Interventions: Other: Nasometry

INTERVENTIONS:
Other: Nasometry — Repetition of several stimuli (syllables, sentences ) in the microphones of the Nasometer

SUMMARY:
The velopharyngeal mechanisms (in particular the movements of the soft palate) is frequently affected by craniofacial anomalies such as cleft lip and palate. Nasofibroscopy is frequently used in clinical care to assess the velopharyngeal function because it allows for direct visualization of the velopharyngeal port. However, it is an invasive procedure that could not be tolerated well by children.

Nasometry is a non-invasive acoustic measurement technique which can be used to objectively assess a velopharyngeal dysfunction (whether it can be heard or not), and thus supplement the perceptual evaluation conducted by a trained clinician.

The main objective of this study is to establish normative nasalance scores with the KayPENTAX Nasometer (Nasometer II 6450 model) for native French-speaking children between 8 and 10 years old.

DETAILED DESCRIPTION:
The velopharyngeal mechanism (in particular the movements of the soft palate) is frequently affected by craniofacial anomalies such as cleft lip and palate and it needs to be assessed. Indeed, the velopharyngeal sphincter has to be efficient in order to properly isolate the oral cavity from the nasal cavity. Thus, the nasal cavity is protected during swallowing (preventing food or liquids from passing through the nose). It also ensures a correct phonation and articulation of oral phonemes.

A perceptual evaluation of the velopharyngeal function is always conducted by a clinician. But it is a subjective assessment which may need to be supplemented by an objective instrumental assessment. Nasofibroscopy is frequently used in clinical care to evaluate the velopharyngeal function because it allows for direct visualization of the velopharyngeal port. However, it is an invasive procedure that could not be tolerated well by children.

Nasometry on the other hand is a non-invasive acoustic measurement technique. It is based on the relation between nasal and oral acoustic energy and determines a nasalance score. Calculated in real time during speech production, the nasalance is a measure expressed as a percentage : (nasal acoustic energy) / (sum of oral and nasal acoustic energy). The device computing the nasalance score is called a Nasometer.

Thus, in addition to the speech therapist's perceptual evaluation, nasometry can be used to objectively assess and quantify a velopharyngeal dysfunction whether it can be heard or not. However in order to determine if a patient's nasalance score is pathological or not, it must be compared to standardized norms. Yet presently, there are no normative nasalance data for French-speaking children. The main objective of this study is to establish normative nasalance scores with the KayPENTAX Nasometer (Nasometer II 6450 model) for native French-speaking children between 8 and 10 years old.

ELIGIBILITY:
Inclusion Criteria:

* Holders of parental authority and patients informed and not opposing their participation in the study
* Patients aged 8 to 10 years old
* native-French speakers (French from France including the French overseas departments and territories)
* Educated in France in an ordinary environment
* Patients without a cleft
* Patients with a cleft : patients with a hard and/or soft palate cleft and for whom the perceptual speech-language pathology evaluation revealed a velopharyngeal insufficiency

Exclusion Criteria:

Patients without developmental speech disorder (including articulation disorder) or hearing impairment

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the Pediatric ENT department of Necker-Enfants Malades hospital
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Nasalance score for each stimulus | Day 0
  Average value of nasalance score for each stimulus
Nasalance score per context | Day 0
  Average value of nasalance score per context (oral - nasal)
Nasalance score of the nasalance distance | Day 0
  Average value of the nasalance distance (difference between the average in a nasal context and the average in an oral context)

SECONDARY OUTCOMES:
Effect of the context on the nasalance scores | Day 0
  Effect of the context (oral / nasal) on the nasalance scores: comparison of the mean, minimum and maximum measurements between the two contexts
Speech stimulus length effect on the nasalance scores | Day 0
  Check whether there is a speech stimulus length effect: are the nasalance scores comparable between repeating an oral short sentence and an oral long sentence, provided that the phonemic distribution is identical? Comparison of the average, minimum and maximum scores between the two stimuli
Effect of the phonetic context on the nasalance scores | Day 0
  Check if there is an effect of the phonetic context (types of vowels and consonants) on the nasalance scores: comparison of the mean, minimum and maximum scores between for example high vowels ([i]) and low ([a]) or between voiceless ([k]) and voiced ([g]) consonants
Test-retest reliability of the nasalance scores | Day 0
  Evaluate the test-retest reliability: selection of a few subjects who will repeat the stimuli twice. Analyze if there is a significant difference between the two repetitions
Most relevant stimuli for a nasometric protocol | Day 0
  Validate the nasometric evaluation protocol for its clinical use : on the basis of speech therapy assessment results, determine the best time / efficiency ratio and choose the most relevant stimuli in order to have the maximum information in a minimum of time
Analysis of acoustic signals captured by standard microphones | Day 0
  Compare the nasalance score obtained with the Nasometer with a nasalance score calculated on the basis of acoustic signals captured at the same time by standard microphones placed on the Nasometer plate: compare the average, minimum and maximum values between the two recordings of acoustic signals

CONTACTS AND LOCATIONS:
Overall Officials: Natacha KADLUB, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Cécile CHAPUIS-VANDENBOGAERDE, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbier H, Redouloux L, Chapuis-Vandenbogaerde C, Picard A, Amelot A, Fougeron C, Sanquer E, Kadlub N. Normative data on nasalance scores for French speaking children. J Stomatol Oral Maxillofac Surg. 2025 Jun;126(3):102089. doi: 10.1016/j.jormas.2024.102089. Epub 2024 Sep 21. PMID 39313155